CLINICAL TRIAL: NCT01635426
Title: Aspirin Versus Clopidogrel Effect on Uterine Perfusion in Women With Unexplained Recurrent Pregnancy Loss With Decreased Uterine Artery Pulsatility Index: A Randomized Controlled Trial
Brief Title: Aspirin Versus Clopidogrel Effect on Uterine Blood Flow in Women With Unexplained Recurrent Miscarriages
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed Ellaithy, Lecturer of Obstetrics & Gynecology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASUOGRCT976
Record Dates: First submitted 2012-07-04; First posted 2012-07-09 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Recurrent Pregnancy Loss
Keywords: Aspirin; Clopidogrel; Unexplained recurrent pregnancy loss; Uterine artery pulsatility index
MeSH Terms: interventions — Aspirin; Clopidogrel

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aspirin (Active Comparator)
  Interventions: Drug: Aspirin
- Clopidogrel (Active Comparator)
  Interventions: Drug: Clopidogrel

INTERVENTIONS:
Drug: Aspirin — Aspirin 75 mg daily for 2 months after meals
  Other Names: Acetylsalicylic Acid
  Arms: Aspirin
Drug: Clopidogrel — Clopidogrel 75 mg daily for 2 months after meals
  Other Names: Plavix
  Arms: Clopidogrel

SUMMARY:
The study will compare the effect of Aspirin versus clopidogrel effect on uterine perfusion in women with unexplained recurrent pregnancy loss with decreased uterine artery pulsatility index.

Null hypothesis: Women with recurrent miscarriage have the same blood flow after aspirin or clopidogrel treatment compared to their uterine artery pulsatility index before treatment.

DETAILED DESCRIPTION:
Recurrent miscarriage has been associated with genetic, anatomic, endocrine, immunologic, behavioral, environmental factors and prothrombotic states; however, almost 50% of cases of recurrent miscarriage are unexplained.

Angiogenesis and uterine blood supply are essential for both endometrial growth and embryo development. As a result, endometrial vascularity has been considered to play a critical role in endometrial receptivity formation and pregnancy maintenance. The development of three-dimensional (3D) ultra-sonography with power Doppler angiography provides an objective and reproducible way to determine endometrial-subendometrial vascularity , which may evaluate quantitatively the uterine vascularity microenvironment for the developing embryo.

Few studies have shown the application of 3D-power Doppler angiography in assessment of pregnancy loss.

The rationale behind the use of aspirin is that this substance, at low doses, produces a vasodilatatory effect by shifting the TXA2/PGI2 ratio toward the dominance of PGI2 activity through the inhibition of TXA2 production. TXA2 is synthesized mainly by platelets and induces platelet aggregation and vasoconstriction, whereas PGI2, produced at the level of vascular endothelial cells, inhibits platelet aggregation and promotes vasodilatation. Aspirin, at low doses, has been proven to produce the selective inhibition of TXA2 production. In fact, TXA2 is primarily produced by the activity of cyclooxygenase prostaglandin synthase-1 (COX-1) at the platelet level, which is highly sensitive to aspirin inhibition. In contrast, PGI2 is mainly synthesized in the endothelial cells through the activity of both COX-1 and COX-2, which is insensitive to aspirin administration at low doses. Therefore, the administration of aspirin at low doses reduces TXA2 production without affecting PGI2 secretion. It is reasonable that the increased PGI2 vasodilatation activity can enhance uterine perfusion, thereby improving reproductive outcome. In addition, it has been hypothesized that aspirin administration can reduce TXA2 endometrial cell excretion. It is known that TXA2 levels at the site of embryo implantation are crucial for the success of pregnancy. The presence of lower endometrial cell TXA2 production has been demonstrated in patients who became pregnant with respect to those who did not achieve pregnancy. For these reasons, low dose Aspirin supplementation is currently considered as an effective and safe treatment option in the prevention of several pregnancy complications.

Nevertheless, aspirin even when administered at low doses can cause gastrointestinal bleeding, as reported in studies using 30-50 mg daily. In addition, it has not been proved that enteric-coated or buffered aspirin is less likely to cause gastrointestinal bleeding than normal aspirin.

The search for active anti-platelet drugs within the original chemical class of the thienopyridines, led to the discovery of clopidogrel, a novel ADP-selective agent whose anti-aggregating properties are several times higher than those of ticlopidine. The anti-aggregating properties of this compound are well known and, very recently, new results have clarified its mechanism of action.

Clopidogrel is active only after intravenous or oral administration, and no circulating activity has been found in the plasma of treated animals or human volunteers.

Experiments in rats have demonstrated that the anti-aggregating activity was caused by a short lasting metabolite generated in the liver by a cytochrome P450-dependent pathway. The anti-aggregating property of clopidogrel is caused by an inhibition of the binding of ADP to its platelet receptors, and more specifically to the low affinity receptors, the high affinity binding sites being unaffected by clopidogrel. Several events in the ADP activation process, including adenylyl cyclase down-regulation, protein tyrosine phosphorylation, activation of the GPIIb-IIIa complex, fibrinogen binding, aggregation and release, were inhibited by clopidogrel and indicate their close relationship with the activation of a low affinity receptor by ADP. Thus, clopidogrel is not only a potent antithrombotic drug in humans but also a good tool to study the effect of ADP on platelets.

The purpose of this study is to compare the effect of Aspirin versus clopidogrel effect on uterine perfusion in women with unexplained recurrent pregnancy loss with decreased uterine artery pulsatility index.

ELIGIBILITY:
Inclusion Criteria:

* Women aged between 20 to 38 years old.
* Regular menstrual cycle (26 to 33 days).
* Women with 2 or more previous unexplained first trimester miscarriage.
* Impaired uterine perfusion (PI of uterine artery more than 2.5).

Exclusion Criteria:

* Known hypersensitivity to any of study medication components.
* Immunotherapy, endocrinotherapy, anticoagulant or anti-platelet management during the past 3 months

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2012-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Improvement in uterine artery pulsatility index | 2 months

SECONDARY OUTCOMES:
Improvement in subendometrial blood flow | 2 month

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Ellaithy, M.D., Principal Investigator — Ain Shams University
Locations (1):
- Ain Shams University, Al ‘Abbāsīyah, Cairo Governorate, Egypt